CLINICAL TRIAL: NCT02068183
Title: Early Identification of World Trade Center Conditions in Adolescents
Brief Title: World Trade Center Adolescent Health Study
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: S12-03116; U01OH010394 (NIH)
Record Dates: First submitted 2014-01-22; First posted 2014-02-21 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Asthma; Hypertension; Cardiovascular Risk Factor; Insulin Resistance; Stress Disorders, Post-Traumatic; Exposure to Toxic Dust
Keywords: World Trade Center exposure; cardiovascular risk; insulin resistance; post-traumatic stress; pulmonary disease
MeSH Terms: conditions — Asthma; Hypertension; Insulin Resistance; Stress Disorders, Post-Traumatic; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — A research assistant well trained in pediatric phlebotomy will collect 25 mL of blood at the first visit, as one aliquot of 3 ml blood in a lavender top vacutainer for CBC, one aliquot of 5 ml blood in a goldtop vacutainer for whole blood, and one 3 ml of blood in a PAX Gene (PreAnalitycX - Hombrechtikon, Switzerland) tube for RNA isolation. One 4 ml cryovial of whole blood will be reserved for future DNA analysis and heavy metal analysis, and another 10 ml vacutainer will be reserved for persistent organic pollutants, while the blood in the PAX Gene will be stored for RNA isolation.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- World Trade Center exposed group: After informed consent, anthropometric and blood pressure/brachial artery distensibility assessments; physical examination and environmental and respiratory history questionnaire completion; heart rate variability measurement; and spirometry/IOS will be performed on the World Trade Center exposed group. A research assistant well trained in pediatric phlebotomy will collect 23 mL of fasting blood. Spirometry and IOS, diet diary collection, lung volumes by plethysmography, and arterial wall stiffness.
- Unexposed comparison group: After informed consent, anthropometric and blood pressure/brachial artery distensibility assessments; physical examination and environmental and respiratory history questionnaire completion; heart rate variability measurement; and spirometry/IOS will be performed on the unexposed comparison group. A research assistant well trained in pediatric phlebotomy will collect 23 mL of fasting blood. Spirometry and IOS, diet diary collection, lung volumes by plethysmography, and arterial wall stiffness.

SUMMARY:
The proposed study builds upon preliminary studies in self-selected populations to identify opportunities for early identification of World Trade Center-related health consequences in adolescents. If adverse health consequences are identified, proactive cardiometabolic and pulmonary screening of exposed children may be indicated, with targeted interventions intended to prevent development of chronic obstructive pulmonary disease, and adverse cardiometabolic outcomes in adulthood.

DETAILED DESCRIPTION:
The study will assess the potential for longer-latency cardiometabolic and pulmonary effects of early life exposure to the World Trade Center (WTC) disaster, and to identify opportunities for early identification of WTC-related health consequences. Preliminary data from the only investigators who regularly provide clinical care to children who lived/attended school near the WTC site identified decrements in spirometry associated with dust cloud exposure, and a remarkably high frequency of cardiometabolic risk factors. Findings from this clinically, self-selected population cannot be extrapolated to the entire population of children who were exposed to the disaster but nonetheless suggest that further study is warranted of the possible metabolic and cardiovascular consequences of WTC exposures. If associated with WTC exposures in a larger, more representative sample, two new and innovative techniques, oscillometry and pulse wave velocity assessment, hold great promise for earlier detection of WTC-related pulmonary and cardiometabolic disease, for whom dietary, environmental and medication interventions may prevent disease progression in later life.

The study will recruit 225 adolescents who respond to the WTC Health Registry (WTCHR), the most representative pediatric population and best-characterized from an environmental exposure standpoint. Connecting the study to the WTCHR also presents efficiency of federal resource utilization, providing more objective clinical data to support self-reported findings of increased persistent respiratory symptoms captured by the WTCHR, thereby improving reliability of the registry data. We will compare pulmonary and cardiometabolic outcomes to carefully matched (age, race/ethnicity, gender, and socioeconomic status) and unexposed control (not resident/attending school south of Houston Street on September 11, 2001) populations from NYU School of Medicine affiliated primary care (private and public clinics).

ELIGIBILITY:
Inclusion Criteria:

* WTCHR participants (exposed group): previous response to WTCHR, born between September 11, 1993 and September 10, 2001
* Controls who are did not live or attend school south of Canal Street on September 11, 2001, matched for age, race/ethnicity, socioeconomic status and other characteristics

Exclusion Criteria:

* Inability to follow procedures.
* Serious lung or heart condition
* Heart or lung surgery
* Uncontrolled asthma
* Current upper respiratory infection
* Pregnancy

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study population for the present proposal will be drawn from the pediatric component of the WTCHR, a cohort of 71,436 adults and children who were first interviewed in 2003-04. To further investigate the associations of WTC exposures with health outcomes, we will compare health parameters in the cohort of WTCHR registrants with 225 subjects in a control cohort drawn from pediatric and adolescent clinics in Manhattan and Brooklyn.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2013-12; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Pulmonary Function Testing | One time
  We will perform spirometry according to standards outlined by the American Thoracic Society and the European Respiratory Society. Specifically, we will assess forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), FEV1/FVC ratio, and forced expiratory flow over 25-75% of the vital capacity (FEF25-75%; Jaeger Masterscreen IOS; Carefusion, Yorba Linda, CA). National Health and Nutrition Examination Survey (NHANES) III reference equations will be used to determine normative values, with statistical analysis to be applied to percents of predicted volumes based on these norms.
Oscillometry | One time
  Oscillometry provides a noninvasive measure of the impedance to airflow within the lung. An externally-generated pressure impulse is applied during tidal breathing in a seated position for 30 seconds, and volume and flow measurements are made.
Plethysmography | One time
  Measured lung volumes will include total lung capacity (TLC), vital capacity (VC), residual volume (RV), and functional residual capacity (FRC) and will be compared to normative values, using established pediatric reference equations.
Blood Pressure | One time
  We will perform assess systolic (first Korotkoff phase) and diastolic (fifth Korotkoff phase) BP three consecutive times in all participants.
Arterial Wall Stiffness | One time
  Pulse Wave Velocity (PWV) will be measured using the SphygmoCor CPV System (AtCor Medical, Sydney, Australia). PWV measures the speed for the pressure wave generated by cardiac ejection to reach the periphery.
Heart Rate Variability | One time
  Assessment of Heart Rate Variability (HRV) will be performed using the SphgymoCor SCOR-CPV device (AtCor Medical, Sydney, Australia).
Insulin resistance | One time
  Fasting insulin and blood glucose will be assessed.

SECONDARY OUTCOMES:
Lipid levels | One time
  Fasting blood draw will be performed.
Psychosocial stress and mental health outcomes | One time
  1. WTC disaster trauma-We will measure psychologically relevant WTC exposure, using questions about direct exposure, family/friend exposure, and media exposure.
  2. Other lifetime trauma
  3. Depression
  4. Substance abuse, and other diagnoses
  5. Post-traumatic stress disorder
  6. Functional impairment
  7. Mental health service utilization
Tobacco smoke exposure | One time
  We will measure tobacco smoke exposure from salivary cotinine.

OTHER OUTCOMES:
Physical activity questionnaire | One time
  Questionnaire adapted from the International Physical Activity Questionnaire-Short last seven days
Diet history questionnaire | One time
  web-based Diet History Questionnaire II developed by the National Cancer Institute

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Trasande, MD, MPP, Principal Investigator — NYU Sch of Med
Locations (1):
- NYU School of Medicine, New York, New York, United States

REFERENCES:
- [Background] Trasande L, Fiorino EK, Attina T, Berger K, Goldring R, Chemtob C, Levy-Carrick N, Shao Y, Liu M, Urbina E, Reibman J. Associations of World Trade Center exposures with pulmonary and cardiometabolic outcomes among children seeking care for health concerns. Sci Total Environ. 2013 Feb 1;444:320-6. doi: 10.1016/j.scitotenv.2012.11.097. Epub 2012 Dec 29. PMID 23280289
- [Derived] Gaylord A, Berger KI, Naidu M, Attina TM, Gilbert J, Koshy TT, Han X, Marmor M, Shao Y, Giusti R, Goldring RM, Kannan K, Trasande L. Serum perfluoroalkyl substances and lung function in adolescents exposed to the World Trade Center disaster. Environ Res. 2019 May;172:266-272. doi: 10.1016/j.envres.2019.02.024. Epub 2019 Feb 16. PMID 30822559
- [Derived] Trye A, Berger KI, Naidu M, Attina TM, Gilbert J, Koshy TT, Han X, Marmor M, Shao Y, Giusti R, Goldring RM, Trasande L. Respiratory Health and Lung Function in Children Exposed to the World Trade Center Disaster. J Pediatr. 2018 Oct;201:134-140.e6. doi: 10.1016/j.jpeds.2018.06.009. Epub 2018 Jul 18. PMID 30029866
- [Derived] Trasande L, Koshy TT, Gilbert J, Burdine LK, Marmor M, Han X, Shao Y, Chemtob C, Attina TM, Urbina EM. Cardiometabolic profiles of adolescents and young adults exposed to the World Trade Center Disaster. Environ Res. 2018 Jan;160:107-114. doi: 10.1016/j.envres.2017.09.026. Epub 2017 Sep 30. PMID 28972913
- [Derived] Koshy TT, Attina TM, Ghassabian A, Gilbert J, Burdine LK, Marmor M, Honda M, Chu DB, Han X, Shao Y, Kannan K, Urbina EM, Trasande L. Serum perfluoroalkyl substances and cardiometabolic consequences in adolescents exposed to the World Trade Center disaster and a matched comparison group. Environ Int. 2017 Dec;109:128-135. doi: 10.1016/j.envint.2017.08.003. Epub 2017 Sep 8. PMID 28890218